CLINICAL TRIAL: NCT06746012
Title: Designing a Dyad-Based MHealth Intervention to Improve Adherence to Lifestyle Recommendations in Colorectal Cancer Survivors and Their Family Caregivers: Human-Centered Study
Brief Title: Designing a Dyad-Based MHealth Intervention to Improve Adherence to Lifestyle Recommendations in Colorectal Cancer Survivors and Their Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Roberto Benzo, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: OSU-23222; NCI-2024-01073 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Stage I Colon Cancer AJCC V8; Stage I Rectal Cancer AJCC V8; Stage II Colon Cancer AJCC V8; Stage II Rectal Cancer AJCC V8; Stage III Colon Cancer AJCC V8; Stage III Rectal Cancer AJCC V8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Interviews as Topic; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (design) (Active Comparator): Survivor-caregiver dyads and SMEs complete semi-structured interview over 60-90 minutes and surveys over 15 minutes for intervention content, format, and feature design and development on study
  Interventions: Other: Survey Administration
- Phase II (user-experience testing) (Active Comparator): Dyads complete semi-structured interview and participate in think-aloud sessions over 60-90 minutes and complete surveys over 15 minutes to test the Healthy Buckeyes app on study.
  Interventions: Procedure: Discussion; Other: Interview; Other: Survey Administration
- Phase III (pilot study) (Experimental): Dyads use the Healthy Buckeyes app to set goals, self-monitor, elicit social support, reinforcement, time management, relapse prevention, and receive exercise videos and recipes tailored to CRC survivors on study. Dyads also watch three 3 minute videos on strategies for improving healthy lifestyle behaviors weekly, wear a Fitbit and use exercise bands, and receive health coaching over 10 weeks on study. Dyads will be prompted through the app to identify specific ways they will support each other (team activity and team huddle) in meeting their goals throughout the week for 10 weeks on study.
  Interventions: Other: Educational Activity; Other: Internet-Based Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Supportive Care; Other: Survey Administration

INTERVENTIONS:
Procedure: Discussion — Participate in think-aloud sessions
  Other Names: Discuss
  Arms: Phase II (user-experience testing)
Other: Educational Activity — Receive health coaching
  Arms: Phase III (pilot study)
Other: Internet-Based Intervention — Use Healthy Buckeyes app
  Arms: Phase III (pilot study)
Other: Internet-Based Intervention — Watch videos
  Arms: Phase III (pilot study)
Other: Interview — Complete semi-structured interview
  Arms: Phase II (user-experience testing); Phase III (pilot study)
Other: Medical Device Usage and Evaluation — Wear Fitbiit and use exercise bands
  Arms: Phase III (pilot study)
Other: Questionnaire Administration — Ancillary studies
  Arms: Phase III (pilot study)
Other: Supportive Care — Receive caregiver support
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Phase III (pilot study)
Other: Survey Administration — Complete surveys

SUMMARY:
This clinical trial develops and tests a mobile health (mHealth) intervention to improve adherence to lifestyle recommendations in colorectal cancer (CRC) survivors and their family caregivers. The current challenge for cancer survivorship is identifying novel approaches to help adhere to the lifestyle recommendations that have been shown to improve symptom burden, health outcomes, and health-related quality of life (HRQoL). The development of a digital health intervention specifically for CRC survivors and family caregivers may improve adherence to the American Cancer Society Nutrition and Physical Activity Guideline for Cancer Survivors and improve family health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct semi-structured interviews with 12 CRC survivors, 12 family caregivers, and 12 subject matter experts (SMEs) to assess the needs, contexts, and perspectives to improve engagement application (app).

II. Develop iterations of a working prototype app by collecting user feedback via semi-structured interviews, think-aloud sessions, and surveys in 12 survivors and 12 caregivers.

III. Conduct a 12-week, single-arm pilot study to test the digital lifestyle intervention's acceptability, feasibility, and intended effects in 10 CRC survivors-caregiver dyads.

OUTLINE:

PHASE I (DESIGN): Survivor-caregiver dyads and SMEs complete semi-structured interview over 60-90 minutes and surveys over 15 minutes for intervention content, format, and feature design and development on study

PHASE II (USER-EXPERIENCE TESTING): Dyads complete semi-structured interview and participate in think-aloud sessions over 60-90 minutes and complete surveys over 15 minutes to test the Healthy Buckeyes app on study.

PHASE III (PILOT STUDY): Dyads use the Healthy Buckeyes app to set goals, self-monitor, elicit social support, reinforcement, time management, relapse prevention, and receive exercise videos and recipes tailored to CRC survivors on study. Dyads also watch three 3 minute videos on strategies for improving healthy lifestyle behaviors weekly, wear a Fitbit and use exercise bands, and receive health coaching over 10 weeks on study. Dyads will be prompted through the app to identify specific ways they will support each other (team activity and team huddle) in meeting their goals throughout the week for 10 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS INCLUSION:
* Adults (18 years of age or older)
* Diagnosis of stage I-III colon or rectal cancer
* Undergone curative-intent complete surgical resection (patients who have received non-operative management for rectal cancer may be eligible)
* Completed treatment (i.e., neo-adjuvant, adjuvant cytotoxic chemotherapy, radiation, or surgical resection) at least six months prior
* Own a smartphone with internet access and can receive text messages
* Able to speak, read, and understand English
* Self-report ability to independently engage in physical activity determined by the Physical Activity Readiness questionnaire (PAR-Q), and if indicated obtain physician clearance
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 determined via medical chart review
* Presence of a family caregiver (i.e., informal or formal caregiver) willing support the patient and participate in the study
* Able to provide informed consent
* FAMILY CAREGIVER INCLUSION:
* Any adult that resides in the same household as the patient
* Willing to participate in all aspects of the intervention and in the assessments required for those in the wait-list control condition if applicable
* Meets the patient inclusion criteria number 1, 5, 6, and 10
* SMES INCLUSION:
* Medical, radiation, and surgical oncologists; advanced practice providers, registered nurses; dietitians; exercise physiologists; physical therapists, patient navigators and champions/advocates, and social workers with at least 12 months of experience working with CRC survivors

Exclusion Criteria:

* PATIENTS EXCLUSION:
* People with potential contraindications to exercise based on the PAR-Q, for those we are unable to obtain physician clearance
* Planned major surgery during the study period
* Scheduled to receive any form of cancer therapy during study participation
* Concurrent, actively treated other cancer (except non-melanoma skin cancer, in situ cervical cancer or localized prostate cancer treated with surveillance only)
* Self-reported history of severe cardiovascular, respiratory, musculoskeletal disease, or joints problems that preclude moderate physical activity (PA)
* Self-reported history of psychiatric disorders that preclude participation in the study intervention or prevent the patient from giving informed consent
* Concurrent participation in another weight loss, PA, or dietary intervention clinical trial
* Currently pregnant or trying to become pregnant during the study period
* living outside the United States (US) during the study period
* Currently a prisoner
* FAMILY CAREGIVER EXCLUSION:
* The same as the patient exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived usability (Phase II) | Up to 1 year
  Will be evaluated via the System Usability Scale (SUS), a ten-item questionnaire rated on a 5-point Likert scale, with a high level of reliability with a coefficient alpha of 0.91.
End user's perception of the quality of the mHealth application (Phase II) | Up to 1 year
  Will be assessed using the User Mobile Application Rating Scale (uMARS), which includes 20 items rated on a 5-point scale and a total of six sections, including engagement, functionality, aesthetics, information quality, subjective quality, and perceived impact.
User acceptance of mHealth services (Phase II) | Up to 1 year
  Will be assessed using the Technology Acceptance Model (TAM), which displays how users use and accept technology. The TAM includes 12 items divided into perceived usefulness and perceived ease of use.
Usability (Phase III) | Up to 1 year
  Will be assessed using the SUS, a 10-item scale, with a score ranging from 0 to 100; where a score of > 68 is considered above average.
Acceptability of the program (Phase III) | Up to 1 year
  Will be determined using the Net Promoter Score (NPS), a single-item 11-point scale asking, "How likely is it that you would recommend to a friend or colleague?" using the NPS survey (Reichheld, 2003). Will deem the program acceptable if the average score is >= 7.
End user's perception of the quality of the mHealth application (Phase III) | Up to 1 year
  Will be assessed using the uMARS (Stoyanov, Hides, Kavanagh, & Wilson, 2016b), which includes 20 items rated on a 5-point scale and a total of six sections, including engagement, functionality, aesthetics, information quality, subjective quality, and perceived impact.
Recruitment rate (Phase III) | Up to 1 year
  Will be defined as the percentage of screened and eligible participants who enroll, and determined 50% as an acceptable threshold.
Adherence rate (Phase III) | Up to 1 year
  Will be defined as the number of participants who used the digital devices as indicated, and determined 70% as an acceptable threshold.
Retention rate (Phase III) | Up to 1 year
  Will be defined as the percentage of enrolled participants who complete the program, and determined 70% as an acceptable threshold.
Acceptability of the measurement rate (Phase III) | Up to 1 year
  Will be defined as the number of participants who complete both the baseline and post-assessment measures.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto M Benzo, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu